CLINICAL TRIAL: NCT02466867
Title: An Open-Label, Multi-Center, Multiple-Application Pharmacokinetic Study of Naftin® (Naftifine Hydrochloride) Cream, 2% in Pediatric Subjects With Tinea Corporis
Brief Title: An Open Label Pharmacokinetic Study of Naftin for Tinea Corporis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Merz North America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MUS90200_4025_1
Record Dates: First submitted 2014-10-29; First posted 2015-06-09 (Estimated); Last update posted 2016-10-28 (Estimated); Status verified 2016-10

CONDITIONS: Tinea Corporis
Keywords: Ringworm
MeSH Terms: conditions — Tinea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Naftin® Cream, 2% (younger pediatric cohort) (Experimental): Subject aged 2 years to 5 years, 11 months with tinea corporis
  Interventions: Drug: Naftin® Cream, 2% (younger pediatric cohort)
- Naftin® Cream, 2% (older pediatric cohort) (Experimental): Subject aged 6 years to 11 years, 11 months with tinea corporis
  Interventions: Drug: Naftin® Cream, 2% (older pediatric cohort)

INTERVENTIONS:
Drug: Naftin® Cream, 2% (younger pediatric cohort) — Approximately 3 grams of Naftin® Cream, 2% ist to be applied once per day for subjects aged 2 to 5 years, 11 months.
  Arms: Naftin® Cream, 2% (younger pediatric cohort)
Drug: Naftin® Cream, 2% (older pediatric cohort) — Approximately 4 grams of Naftin® Cream, 2% ist to be applied once per day for subjects aged 6 to 11 years, 11 months.
  Arms: Naftin® Cream, 2% (older pediatric cohort)

SUMMARY:
This is an open label, multi-center, multi-application pharmacokinetic study in pediatric subjects with tinea corporis.

ELIGIBILITY:
Inclusion Criteria:

* Male or females 2 to 11 years, 11 months of any race. Females of child producing age (started menarche) must have a negative urine pregnancy test.
* Presence of tinea corporis characterized by clinical evidence of a tinea infection at multiple sites covering a total of at least 1% body surface area.
* KOH positive and culture positive baseline skin scrapings obtained from the site most severely affected of the overall severity.
* Subjects must be in good health and free from clinically significant disease that might interfere with the study evaluations.

Exclusion Criteria:

* Tinea infection of the scalp, face, groin, and/or feet.
* A life-threatening condition (ex. autoimmune deficiency syndrome, cancer) within the last 6 months
* Subject with abnormal findings-physically or laboratory- that considered by the investigator to be clinically important and indicative of conditions that might complicate interpretation of study results.
* Subjects with a known hypersensitivity or other contradictions to study medications or their components.

Ages: 2 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 27 (Actual)
Dates: Start 2014-01; Primary Completion 2015-10 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
To quantify the plasma concentration of single and multiple dose of naftifine hydrochloride cream, 2% in pediatric subjects with tinea corporis | 2 weeks
  AUC0-24, Cmax, AUC0-24/D, Cmax/D, AUCt,ss, Cmax,ss, AUCt,,ss/D, Cmax,ss/D

SECONDARY OUTCOMES:
Evaluate plasma PK single and multiple dose PK variables | 2 weeks
  tmax and tmax,ss
Evaluate trough plasma PK concentration | 2 weeks
  Ctrough, ttrough,max, Ctrough,max
Evaluate urine PK single and multiple dose variables | 2 weeks
  Ae0-24, fe, CLR, AEt,ss

CONTACTS AND LOCATIONS:
Overall Officials: Alan B. Fleischer, MD, Study Director — Merz North America, Inc.
Locations (3):
- Merz Investigative Site#001261, College Station, Texas, United States
- Merz Investigative Site#180001, Santo Domingo, Dominican Republic
- Merz Investigative Site #504001, San Pedro Sula, Honduras